CLINICAL TRIAL: NCT00626548
Title: A Phase III, Randomised, Placebo-controlled, Double-blind Study to Assess the Efficacy and Safety of Once-daily Orally Administered ZD4054 (Zibotentan) 10 mg in Non-metastatic Hormone-resistant Prostate Cancer Patients
Brief Title: A Phase III Trial of ZD4054 (Zibotentan) (Endothelin A Antagonist) in Non-metastatic Hormone Resistant Prostate Cancer
Acronym: ENTHUSE M0
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: early efficacy review by the Independent Data Monitoring Committee indicated it was unlikely to meet its primary efficacy endpoints
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4320C00015
Record Dates: First submitted 2008-01-24; First posted 2008-02-29 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: Hormone Resistant Prostate Cancer; Endothelin A Receptor Antagonist; Endothelin A; Endothelin A antagonist
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Palcebo
- ZD4054 (Experimental): ZD4054 (Zibotentan)
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: ZD4054 — 10 mg once daily oral dose
  Other Names: Zibotentan
  Arms: ZD4054
Drug: Palcebo — Matching Plcebo oral tablet once daily
  Arms: Placebo

SUMMARY:
Enthuse M0 is a large phase III clinical trial studying the efficacy of ZD4054 (Zibotentan) in hormone resistant prostate cancer (HRPC).

This clinical trial will test if the Endothelin A Receptor Antagonist ZD4054 (Zibotentan) can improve progression-free survival and overall survival against a background of existing prostate cancer treatments.

ZD4054 (Zibotentan) is a new type of agent, which is thought to slow tumour growth and spread by blocking Endothelin receptor activity. This trial will look at the effects of ZD4054 (Zibotentan) in hormone resistant prostate cancer (HRPC) patients who have had rising PSA after surgical or medical castration but have no evidence of metastases.

All patients participating in this clinical trial will receive existing prostate cancer treatments in addition to trial therapy.

Half the patients will receive ZD4054 (Zibotentan) , and half the patients will receive placebo in addition to standard prostate cancer therapy. By participating in this trial there is a 50% chance that patients will receive an agent that may slow the progression of the tumour.

No patients will be deprived of standard prostate cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients who answer TRUE to the following criteria may be eligible to participate in this study.

* Confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate) that has NOT spread to the other parts of the body (metastases). Patients with lymph node involvement may be eligible if specified criteria is met.
* Increasing Prostate Specific Antigen (PSA), collected within one year of enrollment
* Currently receiving treatment with surgical or medical castration

Exclusion Criteria:

Patients who answer TRUE to the following may NOT be eligible to participate in this study.

* Currently using opiate based pain killers for cancer related pain
* Previous treatment with chemotherapy (paclitaxel, docetaxel, and mitoxantrone). Prior targeted cancer therapies are permitted if received during a previous clinical trial
* Suffering from heart failure or had a myocardial infarction within last 6 months
* A history of epilepsy or seizures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2577 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Miller, Prof., M.D., Principal Investigator — Charite University, Berlin, Germany; Tia Higano, MD, Principal Investigator — University of Washington
Locations (322):
- United States (38):
  - Research Site, Tucson, Arizona
  - Research Site, Greenbrae, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Denver, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Kansas City, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Mystle Beach, South Carolina
  - Research Site, Raleigh, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Seattle, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Santa Fe, Santa Fe Province
- Australia (7):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Hornsby, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Wodonga, Victoria
  - Research Site, Nedlands, Western Australia
  - Research Site, Sydney
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Wels
- Belgium (7):
  - Research Site, (Wilrijk) Antwerpen
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (8):
  - Research Site, Goiânia, Goiás
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Londrina, Paraná
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Canada (18):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfeild Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Point-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Chile (4):
  - Research Site, La Serena
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (11):
  - Research Site, Nanjing, Jiangsu
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hubei
  - Research Site, Jiangsu
  - Research Site, Shanghai
  - Research Site, Shanxi
  - Research Site, Tianjin
  - Research Site, Zejiang
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Medellín
- Czechia (7):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jablonec nad Nisou
  - Research Site, Kroměříž
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Frederiksberg
  - Research Site, Herlev
  - Research Site, Holstebro
  - Research Site, Odense
  - Research Site, Roskilde
- Finland (5):
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, Oulu
  - Research Site, Seinäjoki
  - Research Site, Tampere
- France (17):
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Suresnes
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (26):
  - Research Site, Augsburg
  - Research Site, Bad Ems
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Borken
  - Research Site, Chemnitz
  - Research Site, Emmendingen
  - Research Site, Fürth
  - Research Site, Gelsenkirchen-Buer
  - Research Site, Germering
  - Research Site, Göttingen
  - Research Site, Holzminden
  - Research Site, Kirchheim/Teck
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Mannheim
  - Research Site, Muehlheim An Der Ruhr
  - Research Site, Muenchen-Planegg
  - Research Site, Mühlacker
  - Research Site, München
  - Research Site, Münster
  - Research Site, Reutlingen
  - Research Site, Rostock
  - Research Site, Tübingen
  - Research Site, Waltshut-Tiengen
  - Research Site, Wuppertal
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Székesfehérvár
- India (8):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Nadiād, Gujarat
  - Research Site, Kochi, Kerala
  - Research Site, Pune, Maharashtra
  - Research Site, Chennai, Tamil Nadu, India
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Kolkota, West Bengal
  - Research Site, New Delhi
- Research Site, Dublin, Ireland
- Israel (7):
  - Research Site, Beersheba
  - Research Site, Be’er Ya‘aqov
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jeruslaem
  - Research Site, Petah Tikva
  - Research Site, Tel-HaShomer - Ramat Gan
- Italy (14):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Como
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Rome
  - Research Site, Terni
  - Research Site, Varese
- Japan (35):
  - Research Site, Hirosaki, Aomori
  - Research Site, Chiba, Chiba
  - Research Site, Narashino, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Maebashi, Gunma
  - Research Site, Ōtake, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Ibaraki-machi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kita-gun, Kagawa-ken
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Kamigyō-ku, Kyoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Ueda, Nagano
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Kashihara, Nara
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Osaka, Osaka
  - Research Site, Ōsaka-sayama, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Wako, Saitama
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Fuchu_city, Tokyo
  - Research Site, Itabashi-Ku, Tokyo
  - Research Site, Meguro-ku, Tokyo
  - Research Site, Minato-Ku, Tokyo
  - Research Site, Mitaka, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
- Latvia (2):
  - Research Site, Liepāja
  - Research Site, Riga
- Mexico (2):
  - Research Site, Distrito Federal, Mexico City
  - Research Site, Mexico City, Mexico City
- Netherlands (7):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Eindhoven
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Tilburg
- Norway (2):
  - Research Site, Trondheim
  - Research Site, Tønsberg
- Peru (4):
  - Research Site, Arequipa
  - Research Site, Bellavista
  - Research Site, Jesus Maria
  - Research Site, Lima
- Poland (6):
  - Research Site, Gdynia
  - Research Site, Kielce
  - Research Site, Kościerzyna
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (2):
  - Research Site, Coimbra
  - Research Site, Porto
- Romania (3):
  - Research Site, Timișoara, Timiș County
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Russia (9):
  - Research Site, Omsk, Omsk Oblast
  - Research Site, Izhevsk, Russia
  - Research Site, Tomsk, Tomsk Oblast
  - Research Site, Barnaul
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Voronezh
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Niš
  - Research Site, Novi Sad
- South Africa (6):
  - Research Site, Observatory, Cape Town
  - Research Site, Tygerberg, Cape Town
  - Research Site, Overport, Durban
  - Research Site, Parktown, Johannesburg
  - Research Site, Pietermaritzburg
  - Research Site, Pretoria
- South Korea (6):
  - Research Site, Seo-gu, Busan
  - Research Site, Bundang-Gu, Seongnam-si, Gyeonggi-do
  - Research Site, Gangnam-gu, Seoul
  - Research Site, Seodaemun-gu, Seoul
  - Research Site, Seongbuk-gu, Seoul
  - Research Site, Songpa-gu, Seoul
- Spain (8):
  - Research Site, Elche, Alicante
  - Research Site, Barakaldo, Bizkaia
  - Research Site, Bilbao, Vizcaya
  - Research Site, A Corunna
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Jönköping
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Uppsala
- Switzerland (4):
  - Research Site, Aarau
  - Research Site, Ch-4031 Basel
  - Research Site, Locarno
  - Research Site, Zurich
- Research Site, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (13):
  - Research Site, Reading, Berkshire
  - Research Site, Cottingham, East Yorkshire
  - Research Site, Stevenage, Hertfordshire
  - Research Site, Maidstone, Kent
  - Research Site, Guildford, Surrey
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Huddersfield
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2577 patients with hormone-resistant prostate cancer patients and bone metastasis were recruited between 15th January 2008 and 3rd May 2011
Pre-assignment Details: 1156 of the 2577 enrolled patients were not randomised to treatment groups as they failed screening
Groups:
- ZD4054: ZD4054 10 mg oral tablet once daily
- Placebo: Placebo oral tablet once daily
Period: Overall Study
Arm/Group | ZD4054 | Placebo
Started | 705 | 716
Patients Received Treatment | 703 | 712
Completed | 0 | 0
Not Completed | 705 | 716
Not completed — Adverse Event | 164 | 44
Not completed — Withdrawal by Subject | 42 | 46
Not completed — Protocol Violation | 4 | 11
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other termination reason | 493 | 613

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZD4054 | Placebo | Total
Number analyzed (Participants) | 705 | 716 | 1421
Age Continuous [Mean (Standard Deviation); unit: years]
  Overall | 72.4 (7.8) | 72.5 (7.8) | 72.45 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 705 | 716 | 1421

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of participants who have died at early analysis data cut off (DCO)
Time Frame: From date of randomization until date of death, assessed up to 33 months
Population: The analysis population only includes patients recruited by the time of the early analysis (1 October 2010)
Measure: Number; unit: Participants
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 592 | 589
Participants | 40 | 39

2. Primary Outcome: Progression Free Survival
Description: Number of participants who have a progression event at the early analysis DCO, where progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline
Time Frame: Participants were followed up for progression every 4 weeks for the first 16 weeks then every 16 weeks
Population: The analysis population only includes patients recruited by the time of the early analysis (1 October 2010)
Measure: Number; unit: Participants
Arm/Group | ZD4054 | Placebo
Number analyzed (Participants) | 592 | 589
Participants | 131 | 162

3. Secondary Outcome: Health Related Quality of Life
Time Frame: Participants were followed up every 4 weeks for the first 16 weeks then every 16 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Time Frame: Participants were followed up every 4 weeks for the first 16 weeks then every 16 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Time to Symptomatic Progression
Time Frame: Participants were followed up every 4 weeks for the first 16 weeks then every 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | ZD4054 | Placebo
Serious Adverse Events (participants affected / at risk) | 148/703 | 138/712
Other Adverse Events (participants affected / at risk) | 531/703 | 392/712
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 (N=703) | Placebo (N=712)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hilar Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 9 | 3
Angina Pectoris (Cardiac disorders) | 1 | 7
Myocardial Infarction (Cardiac disorders) | 5 | 3
Atrial Fibrillation (Cardiac disorders) | 4 | 2
Coronary Artery Disease (Cardiac disorders) | 3 | 0
Acute Myocardial Infarction (Cardiac disorders) | 2 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 2
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 2
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac Disorder (Cardiac disorders) | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Diastolic Dysfunction (Cardiac disorders) | 1 | 0
Hypertensive Cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 1
Prinzmetal Angina (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Congenital Aortic Valve Stenosis (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Macular Hole (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Inguinal Hernia (Gastrointestinal disorders) | 2 | 2
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pneumatosis Intestinalis (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectourethral Fistula (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Oedema Peripheral (General disorders) | 4 | 0
Death (General disorders) | 2 | 1
Pyrexia (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 1
Chest Pain (General disorders) | 1 | 0
Device Dislocation (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Impaired Healing (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Medical Device Complication (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 1 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 1
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 5
Urinary Tract Infection (Infections and infestations) | 2 | 3
Bronchopneumonia (Infections and infestations) | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Chronic Sinusitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Parainfluenzae Virus Infection (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Scrotal Abscess (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Chest Injury (Injury, poisoning and procedural complications) | 0 | 2
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 | 1
Cystitis Radiation (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis Radiation (Injury, poisoning and procedural complications) | 1 | 0
Heat Illness (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Open Fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation Proctopathy (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 0 | 1
International Normalised Ratio Increased (Injury, poisoning and procedural complications) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 2
Diabetic Foot (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign Urinary Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 2 | 0
Transient Ischaemic Attack (Nervous system disorders) | 2 | 1
Brain Stem Stroke (Nervous system disorders) | 1 | 0
Cerebellar Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular Disorder (Nervous system disorders) | 0 | 1
Cerebrovascular Insufficiency (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 7
Renal Failure Acute (Renal and urinary disorders) | 5 | 2
Calculus Ureteric (Renal and urinary disorders) | 3 | 0
Renal Failure (Renal and urinary disorders) | 2 | 3
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 2
Renal Impairment (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder Stenosis (Renal and urinary disorders) | 0 | 1
Calculus Bladder (Renal and urinary disorders) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 1
Renal Disorder (Renal and urinary disorders) | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Calculus Prostatic (Reproductive system and breast disorders) | 1 | 0
Pelvic Haematoma (Reproductive system and breast disorders) | 1 | 0
Prostatic Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Peau D'orange (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 2 | 3
Aortic Aneurysm (Vascular disorders) | 0 | 1
Arterial Stenosis (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 0 | 1
Femoral Arterial Stenosis (Vascular disorders) | 1 | 0
Iliac Artery Occlusion (Vascular disorders) | 0 | 1
Intermittent Claudication (Vascular disorders) | 0 | 1
Temporal Arteritis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
twqVenous Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 (N=703) | Placebo (N=712)
Anaemia (Blood and lymphatic system disorders) | 46 | 23
Constipation (Gastrointestinal disorders) | 64 | 76
Diarrhoea (Gastrointestinal disorders) | 46 | 63
Nausea (Gastrointestinal disorders) | 59 | 61
Oedema Peripheral (General disorders) | 268 | 88
Fatigue (General disorders) | 71 | 79
Asthenia (General disorders) | 35 | 43
Rhinitis (Infections and infestations) | 56 | 17
Urinary Tract Infection (Infections and infestations) | 43 | 54
Nasopharyngitis (Infections and infestations) | 34 | 45
Decreased Appetite (Metabolism and nutrition disorders) | 40 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 54
Back Pain (Musculoskeletal and connective tissue disorders) | 33 | 49
Headache (Nervous system disorders) | 188 | 82
Dizziness (Nervous system disorders) | 46 | 39
Haematuria (Renal and urinary disorders) | 23 | 36
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 176 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 33
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 48 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
3. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

AstraZeneca can review results communications prior to public release and may within 60 days of receipt require amendments to be made. AstraZeneca can also require that submission or disclosure be delayed to allow for